CLINICAL TRIAL: NCT03264690
Title: A Prospective Study to Observe the Change in Microbiome in Human Derived Sample and the Relation With Clinical Response Before and After the Anti-TNF Treatment in IBD Patients
Brief Title: Study to Observe the Change in Microbiome in Human Derived Sample and the Relation With Clinical Response Before and After the Anti-TNF Treatment in IBD Patients
Acronym: ETERNITY
Status: Completed | Type: Observational
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: D2E7-M082-602
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2019-11

CONDITIONS: Inflammatory Bowel Disease
Keywords: Crohn's disease; Ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Microbial composition measured from IBD and non-IBD groups: Participants with inflammatory bowel disease (IBD) and non-IBD will be measured for microbial composition.

SUMMARY:
This study will be conducted to observe the difference in microbiome composition between healthy participants and inflammatory bowel disease (IBD) participants with no anti-tumor necrosis factor (anti-TNF) treatment.

ELIGIBILITY:
1. Inclusion/ Exclusion Criteria:

   1. Inclusion Criteria For Inflammatory Bowel Disease (IBD) participants:

      * Male or female, age ≥ 19 years at the time of informed consent
      * Confirmed diagnosis of IBD
      * Participants who are naïve to anti-tumour necrosis factor (anti-TNF)
   2. Exclusion Criteria for IBD participants:

      * Contraindication to anti-TNF including active tuberculosis (TB), sepsis, or other severe opportunistic infection, etc.
2. Inclusion/ Exclusion Criteria:

   1. Inclusion Criteria for non-IBD participants:

      * Participants who have not been diagnosed with IBD
      * Participants who don't have any other intestinal disease except IBD
      * Participants who are naïve to anti-TNF
   2. Exclusion Criteria for non-IBD participants:

      * Participants who have been on medication to treat underlying disease for the previous 3 months

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female participants diagnosed with inflammatory bowel disease (IBD) will be compared to participants with non-IBD.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Change in the composition of the microbiome after anti-tumour necrosis factor (anti-TNF) treatment for inflammatory bowel disease (IBD) at Month 3 | Month 3
  Microbiome is the microorganisms in a particular environment (including the body or a part of the body). Changes in the microbiome in fecal, blood, saliva, and urine samples before and after anti-TNF treatment will be assessed.

SECONDARY OUTCOMES:
The difference in the composition of the microbiome at baseline between IBD participants and non-IBD participants | Baseline
  Microbiome is the microorganisms in a particular environment (including the body or a part of the body). Changes in the microbiome in fecal, blood, saliva, and urine samples before and after anti-TNF treatment will be assessed.
Disease activity will be assessed by Crohn's Disease Activity Index (CDAI) or Mayo score for ulcerative colitis (UC) | Up to 3 months
  Disease activity will be assessed by CDAI to quantify the symptoms.
Correlation in the composition of the microbiome at baseline and disease activity will be assessed as measured by CDAI or Mayo score at Month 3 | Baseline; Month 3
  The composition of the microbiome at baseline will be correlated to disease activity which is assessed as measured by CDAI or Mayo score at Month 3.
Change from baseline in calprotectin at Month 3 | Baseline; Month 3
  Fecal calprotectin can indicate inflammation in the intestines.
Number of participants with abnormal, clinically significant vital signs | Up to 3 months
  Clinical significance will be determined by the investigator.

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Eisai Trial Site # 1, Seoul
  - Eisai Trial Site # 2, Seoul
  - Eisai Trial Site # 3, Seoul